CLINICAL TRIAL: NCT02488850
Title: Determination of Peripheral Immune Cell Activity During Treatment With Either Surgery or Radiotherapy in Patients With Early Stage Non-small Cell Lung Cancer HAMLET Study
Brief Title: Determination of Peripheral Immune Cell Activity During Treatment With Either Surgery or Radiotherapy in Patients With Early Stage NSCLC
Acronym: HAMLET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joachim Aerts, MD PhD, Prof. dr., Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL42081.078.12
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: immune monitoring; T cell activation; early stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

ARMS (2):
- Surgery (Active Comparator): An anatomical surgical resection of primary tumor
  Interventions: Procedure: Surgery
- Radiotherapy (Active Comparator): Stereotactic Ablative Radiotherapy (SABR), outpatient treatment that is typically delivered in between 3-8 fractions
  Interventions: Radiation: SABR

INTERVENTIONS:
Procedure: Surgery
  Arms: Surgery
Radiation: SABR
  Arms: Radiotherapy

SUMMARY:
Rationale: An anatomical surgical resection is considered to be the standard of care in fit patients who present with early stage non-small cell lung cancer (NSCLC). However, surgery is less frequently performed in both elderly patients (aged ≥75 years), who represent the fastest-growing group of patients with stage I/II NSCLC, and in patients who have significant co-morbidity. Following the introduction of stereotactic ablative radiotherapy (SABR), an outpatient treatment that is typically delivered in between 3-8 fractions, the median survival of all elderly patients undergoing radiotherapy in The Netherlands increased by 9.3 months. Randomized trials comparing SABR and surgery have yet to be completed and results of the ongoing ACOSOG Z4032 studies will not be available in the within 5 years. A recent data retrospective study comparing both modalities has raised interesting questions about the impact of local therapy on recurrence patterns. It was found that a better loco-regional disease control rate was achieved with SABR.

Objective: To study the effect of surgery and SABR on both immunostimulatory (with primary endpoint CD8 positive cells) and immunosuppressive cells in peripheral blood in patients with early stage non-small cell lung cancer who are treated with either modality.

Study population: 40 patients with cT1-2aN0M0 either cytologically or histologically proven NSCLC.

Main study parameters/endpoints: To determine whether an increase in CD8 activity can be established after SABR in patients with early stage lung cancer and to compare this increase with that in patients undergoing a surgical intervention. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Only risks in participation are the risks with drawing blood. Subjects will not have any benefits. This pilot study will be used to generate information concerning both treatments useful for the decision to plan a future study in a larger series of patients.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically proven cT1-2aN0M0 NSCLC
* Patients ≥ 18 years old
* Patients should be fit to undergo both treatments in accordance with institutional protocols

Exclusion Criteria:

* Patients with any signs of any co-existing infectious disease or immunosuppressive treatment (inhalation steroids are permitted)
* Mentally incapacitated subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12; Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Number of IFN-gamma/ Granzyme B producing CD8 T cells | Baseline (week 0)
  Number and activation status of peripheral CD8+ T cells
Number of IFN-gamma/ Granzyme B producing CD8 T cells | Week 1
  Number and activation status of peripheral CD8+ T cells
Number of IFN-gamma/ Granzyme B producing CD8 T cells | Week 2
  Number and activation status of peripheral CD8+ T cells
Number of IFN-gamma/ Granzyme B producing CD8 T cells | Week 3
  Number and activation status of peripheral CD8+ T cells
Number of IFN-gamma/ Granzyme B producing CD8 T cells | Week 6
  Number and activation status of peripheral CD8+ T cells

SECONDARY OUTCOMES:
CD4/CD8 ratio in peripheral blood | Baseline
CD4/CD8 ratio in peripheral blood | Week 1
CD4/CD8 ratio in peripheral blood | Week 2
CD4/CD8 ratio in peripheral blood | Week 3
CD4/CD8 ratio in peripheral blood | Week 6
number of regulatory T cells | Baseline
number of regulatory T cells | Week 1
number of regulatory T cells | Week 2
number of regulatory T cells | Week 3
number of regulatory T cells | Week 6
Activation marker expression on T cells | Baseline
Activation marker expression on T cells | Week 1
Activation marker expression on T cells | Week 2
Activation marker expression on T cells | Week 3
Activation marker expression on T cells | Week 6

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Erasmus MC Cancer Institute, Rotterdam, South Holland
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - VU Medical Center, Amsterdam

REFERENCES:
- [Derived] de Goeje PL, Smit EF, Waasdorp C, Schram MTB, Kaijen-Lambers MEH, Bezemer K, de Mol M, Hartemink KJ, Nuyttens JJME, Maat APWM, Hegmans JPJJ, Hendriks RW, Senan S, Aerts JGJV. Stereotactic Ablative Radiotherapy Induces Peripheral T-Cell Activation in Patients with Early-Stage Lung Cancer. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1224-1227. doi: 10.1164/rccm.201610-2178LE. No abstract available. PMID 28345951